CLINICAL TRIAL: NCT01432600
Title: Evaluation of Pomalidomide in Combination With High Dose Dexamethasone and Oral Cyclophosphamide in Patients With Relapsed and Refractory Myeloma
Brief Title: Pomalidomide in Combination With High Dose Dexamethasone and Oral Cyclophosphamide
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16705; PO-MM-PI-0039 (Other Grant/Funding Number: Celgene)
Record Dates: First submitted 2011-09-09; First posted 2011-09-13 (Estimated); Results first posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-02

CONDITIONS: Myeloma
Keywords: Multiple Myeloma; Relapsed; Refractory; Corticosteroids
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma; Recurrence | interventions — pomalidomide; Dexamethasone; Calcium Dobesilate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A: Dose Escalation of Cyclophosphamide (Experimental): Phase I: Pomalidomide, high dose dexamethasone and oral cyclophosphamide:
  Pomalidomide 4 mg by mouth (PO) days 1-21 of a 28 days cycle.
  Dexamethasone 40* mg PO days 1- 4, 15-18 of a 28 days cycle for the first 4 cycles and subsequently 40 mg PO Days 1,8,15, 22. *Participants who were >75 years of age or those who were known to be intolerant to 40 mg weekly dexamethasone received 20 mg dexamethasone on the same schedule.
  Dose Escalation of Cyclophosphamide, orallly (PO) days 1, 8, 15 as follows:
  Level 1: 300 mg; Level 2: 400 mg; Level 3: 500 mg.
  Aspirin 81 mg PO daily (unless the participants had contraindications or were receiving other form of anticoagulation for other indications).
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Cyclophosphamide
- B: Pomalidomide and Dexamethasone (Active Comparator): Randomized Phase II - Pomalidomide high dose dexamethasone:
  Pomalidomide 4 mg PO days 1-21 of a 28 days cycle.
  Dexamethasone 40* mg PO Days 1,8,15, 22. *Participants who were >75 years of age or those who were known to be intolerant to 40 mg weekly dexamethasone received 20 mg dexamethasone on the same schedule.
  Aspirin 81 mg PO daily (unless the participants had contraindications or were receiving other form of anticoagulation for other indications).
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- C: Pomalidomide/Dexamethasone/Cyclophosphamide (Active Comparator): Randomized Phase II - Pomalidomide high dose dexamethasone and oral cyclophosphamide:
  Pomalidomide 4 mg PO days 1-21 of a 28 days cycle.
  Dexamethasone 40* mg PO days 1- 4, 15-18 of a 28 days cycle for the first 4 cycles and subsequently 40 mg PO Days 1,8,15, 22. *Participants who were >75 years of age or those who were known to be intolerant to 40 mg weekly dexamethasone received 20 mg dexamethasone on the same schedule.
  Cyclophosphamide 400 mg PO days 1, 8, 15.
  Aspirin 81 mg PO daily (unless the participants had contraindications or were receiving other form of anticoagulation for other indications).
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Cyclophosphamide
- D: Crossover (Other): Crossover from Arm B to Arm D. Participants who experienced progressive disease in arm B were allowed to crossover to arm D at the discretion of the treating physician, in which case oral weekly Cyclophosphamide (400 mg orally on days 1, 8, and 15) was added to their tolerated dose of pomalidomide and dexamethasone.
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pomalidomide — Pomalidomide at 4 mg by mouth (PO) as outlined in the treatment arms.
  Other Names: CC-4047, POMALYST®
Drug: Dexamethasone — Dexamethasone at 40 mg (20 mg) PO as outlined in the treatment arms.
  Other Names: Decadron®
Drug: Cyclophosphamide — The dose escalation uses a standard "3x3" design: Ex: If none of the first 3 participants have a DLT, enter 3 participants at the next higher dose level. Once the maximum tolerated dose (MTD) of oral weekly cyclophosphamide in combination with pomalidomide and dexamethasone was determined, investigators proceeded with the second phase of the trial, a randomized phase II study comparing pomalidomide and dexamethasone with pomalidomide, dexamethasone and oral weekly cyclophosphamide delivered at the MTD determined in the phase I study.
  Other Names: Cytoxan
  Arms: A: Dose Escalation of Cyclophosphamide; C: Pomalidomide/Dexamethasone/Cyclophosphamide; D: Crossover

SUMMARY:
The main purpose of this study is to see whether pomalidomide can help people with myeloma. Researchers also want to find out if pomalidomide is safe and tolerable.

DETAILED DESCRIPTION:
There are two parts to this study:

* Phase 1: To determine a safe dose of the medication cyclophosphamide in combination with pomalidomide and dexamethasone.
* Phase 2: To see the difference in effectiveness of pomalidomide in combination with high dose dexamethasone with or without cyclophosphamide for the treatment of participants who have myeloma, which has relapsed to or become refractory (not responding) to prior treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have relapsed or refractory multiple myeloma. Refractory disease is defined as patients who experience disease progression on active therapy or within 60 days after the discontinuation of therapy. Relapsed disease is defined as achievement of at least a partial response followed by disease progression after 60 days of discontinuing active therapy.
* Must have measurable disease as assessed by one of the following criteria: Serum monoclonal protein ≥ 0.5 g/dL by protein electrophoresis; >200 mg of monoclonal protein in the urine on 24 hour electrophoresis; Serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
* Must have received at least 2 prior therapies to include prior immunomodulatory drug (lenalidomide) and the patient must be refractory to lenalidomide (defined as progressive disease during active therapy or within 60 days of discontinuation of therapy). All previous cancer chemotherapy (bisphosphonates are not included), including surgery, must have been discontinued ≥2 weeks prior to first dose of study drug. Prior radiotherapy must have been completed > 2 weeks prior to the start of study drug unless the radiation field would not impact marrow reserve in the opinion of the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2 (Karnofsky ≥60%
* Must have acceptable organ function: total bilirubin less than 1.5 mg/dL; aspartic transaminase (AST)/alanine transaminase (ALT) ≤2.5 X institutional upper limit of normal (ULN); serum creatinine < 3mg/dL
* Must have adequate hematologic function as evidenced by the following:
* For the Phase I study: Absolute neutrophil count (ANC) ≥ 1000 per mm³; Platelet count ≥ 50,000 per mm³.
* For the Phase II portion, patients with greater than 50% bone marrow plasmacytosis will be allowed to enter the trial if the platelet count is greater than 30,000 per mm³ and regardless of baseline absolute neutrophil count if it is felt to be related to active myeloma and if in the opinion of the investigator, growth factor support can result in improvement in the neutrophil count to greater than 1000 per mm³ (growth factor can be used during screening).
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy.
* Ability to understand and the willingness to sign a written informed consent document
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid (ASA) may use warfarin or low molecular weight heparin).
* All study participants must be registered into the mandatory POMALYST REMS™ program, and be willing and able to comply with the requirements of the POMALYST REMS™ program.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (see Inclusion Criteria above) or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier (except for neuropathy).
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form
* Any condition, including the presence of laboratory abnormalities, which places the patient at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study. Use of any other experimental drug or therapy within 28 days of baseline.
* Known hypersensitivity to thalidomide or lenalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide, pomalidomide or similar drugs
* Known positive for human immunodeficiency virus (HIV) or infectious hepatitis, type A, B or C
* May not be receiving any other investigational agents
* Pregnant or breast feeding females (Lactating females must agree not to breast feed while taking pomalidomide).
* Patients with prior pomalidomide therapy (greater than 1 cycle) are excluded.
* Another active malignancy requiring treatment within the next 12 months, with the exception of basal cell skin cancer, in situ cervical cancer, in situ breast cancer and asymptomatic prostate cancer
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (except simple urinary tract or upper respiratory tract infection), symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Inability to comply with the protocol requirements or participation in any other clinical study
* Corticosteroid therapies of >20 mg/day prednisone, >4 mg/day dexamethasone, >80 mg/day hydrocortisone, or equivalent
* Allogeneic stem cell/bone marrow transplant within 12 months of first dose of study drug or active graft versus host disease
* Patients with existing peripheral neuropathy grade >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachid Baz, M.D., Principal Investigator — H. Lee Moffitt Cancer and Research Institute
Locations (3):
- United States (3):
  - University of California San Francisco, San Francisco, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Mount Sinai School of Medicine, The Tisch Cancer Institute, New York, New York

REFERENCES:
- [Derived] Baz RC, Martin TG 3rd, Lin HY, Zhao X, Shain KH, Cho HJ, Wolf JL, Mahindra A, Chari A, Sullivan DM, Nardelli LA, Lau K, Alsina M, Jagannath S. Randomized multicenter phase 2 study of pomalidomide, cyclophosphamide, and dexamethasone in relapsed refractory myeloma. Blood. 2016 May 26;127(21):2561-8. doi: 10.1182/blood-2015-11-682518. Epub 2016 Mar 1. PMID 26932802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between December 2011 and March 2014, participants were enrolled at: H. Lee Moffitt Cancer Center and Research Institute, Tampa, FL; UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, CA; Tisch Cancer Institute, Mount Sinai School of Medicine, New York, NY.
Groups:
- A: Dose Escalation of Cyclophosphamide: Phase I: Pomalidomide, high dose dexamethasone and oral cyclophosphamide.
- B: Pomalidomide and Dexamethasone: Phase II: Pomalidomide and high dose dexamethasone.
  Arm D participants may be referenced separately in some Outcome Measures.
- C: Pomalidomide, Dexamethasone, Cyclophosphamide: Phase II: Pomalidomide high dose dexamethasone and oral cyclophosphamide.
Period: Overall Study
Arm/Group | A: Dose Escalation of Cyclophosphamide | B: Pomalidomide and Dexamethasone | C: Pomalidomide, Dexamethasone, Cyclophosphamide
Started | 10 | 36 | 34
Completed | 10 | 35 | 33
Not Completed | 0 | 1 | 1
Not completed — Rapid PD, allocated intv. not rec'd | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants. Arm D (a part of Arm B) started in July 2012 when, per protocol guidelines, 17 participants from Arm B elected to crossover to Arm D. Some measures may include arm D, making the total of participants evaluated higher.
Groups:
- B: Pomalidomide and Dexamethasone: Phase II: Pomalidomide and high dose dexamethasone.
  Crossover Arm D is a part of Arm B. Arm D was opened later to accommodate requested transfers from Arm B. Participants who experienced progressive disease in arm B were allowed to crossover to arm D at the discretion of the treating physician.
  Arm D participants may be referenced separately in some Outcome Measures.
- Total: Total of all reporting groups
Arm/Group | A: Dose Escalation of Cyclophosphamide | B: Pomalidomide and Dexamethasone | C: Pomalidomide, Dexamethasone, Cyclophosphamide | Total
Number analyzed (Participants) | 10 | 36 | 34 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 19 | 17 | 39
  >=65 years | 7 | 17 | 17 | 41
Age, Continuous [Mean (Full Range); unit: years] | 69 [44 to 73] | 64 [50 to 78] | 62 [47 to 80] | 63 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 13 | 16 | 32
  Male | 7 | 23 | 18 | 48
Region of Enrollment [Number; unit: participants]
  United States | 10 | 36 | 34 | 80

OUTCOME MEASURES:

1. Primary Outcome: Phase I - Maximum Tolerated Dose (MTD)
Description: The maximum tolerated dose of oral weekly cyclophosphamide in milligrams (mg), in combination with pomalidomide and dexamethasone. Dose Escalation of Cyclophosphamide, orallly (PO) days 1, 8, 15 as follows: Level 1: 300 mg; Level 2: 400 mg; Level 3: 500 mg. The period for assessment of Dose Limiting Toxicity (DLT) is the first cycle (28 days). The following toxicities will be considered dose limiting if encountered only in the phase I portion of the study: Febrile neutropenia; Grade 3 or 4 non-hematologic toxicity related to treatment with pomalidomide or cyclophosphamide; Participants must have received optimal symptomatic treatment for Grade 3 or 4 nausea, vomiting, or diarrhea to be considered a DLT; Grade 4 transaminitis; Grade 3 transaminitis must be present for ≥ 7 days to be considered a DLT; Grade 4 thrombocytopenia for 7 or more days; Grade 4 neutropenia for 7 or more days.
Time Frame: 28 Days
Population: All Phase I Participants.
Measure: Number; unit: mg
Arm/Group | A: Dose Escalation of Cyclophosphamide
Number analyzed (Participants) | 10
mg | 400

2. Primary Outcome: Phase II - Overall Response Rate (ORR)
Description: Overall response, Minimal Remission (MR) or better per treatment arm, using the uniform response criteria by the International Myeloma Working Group (IMWG) of pomalidomide in combination with high dose dexamethasone with or without cyclophosphamide in participants with relapsed and refractory myeloma. In addition, Minimal response was incorporated in those response criteria as this is a valid endpoint in patients with relapsed or refractory myeloma. MR: 25-49% reduction in serum paraprotein and a 50-89% reduction in urine light chain excretion; A 25-49% reduction in the size of soft tissue plasmacytoma must be demonstrated is applicable.
Time Frame: 36 Months
Population: All Phase II Participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | B: Pomalidomide and Dexamethasone | C: Pomalidomide, Dexamethasone, Cyclophosphamide
Number analyzed (Participants) | 36 | 34
percentage of participants | 38.9 [23 to 54.8] | 64.7 [48.6 to 80.8]

3. Secondary Outcome: Phase II - Median Progression Free Survival (PFS)
Description: Progression free survival per treatment arm. Progressive Disease (PD) requires one of the following, increase of greater than or equal to 25% from baseline in: Serum M-component; Urine M-component; The difference between involved and uninvolved sFLC levels; The size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia.
Time Frame: 36 Months
Population: All Phase II Participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | B: Pomalidomide and Dexamethasone | C: Pomalidomide, Dexamethasone, Cyclophosphamide
Number analyzed (Participants) | 36 | 34
months | 4.4 [2.3 to 5.7] | 9.5 [4.6 to 14]

4. Secondary Outcome: Phase II - Median Overall Survival (OS)
Description: Overall survival per treatment arm. Overall survival is defined as the time from start of treatment to death of any cause.
Time Frame: 36 Months
Population: All participants assigned to Arm B and Arm C.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | B: Pomalidomide and Dexamethasone | C: Pomalidomide, Dexamethasone, Cyclophosphamide
Number analyzed (Participants) | 36 | 34
months | 16.8 [9.3 to NA] — not reached | NA [13.1 to NA] — not reached

5. Secondary Outcome: Phase II - Occurrence of Possibly Related Adverse Events (AEs)
Description: Phase II: Participants with Grade 3 or 4 adverse events at least possibly related to the study treatment in 5% of participants in the Phase 2 portion, by AE category, assessed by the National Cancer Institute Common Terminology Criteria (NCI CTC) version 4.0.
Time Frame: Up to 48 Months
Population: All Phase II Participants who completed allocated intervention.
Measure: Number; unit: percentage of participants
Groups:
- D: Crossover Arm: Phase II: Participants who crossed over from Arm B to Arm D. Crossover Arm D is a part of Arm B. Arm D was opened later to accommodate requested transfers from Arm B. Participants who experienced progressive disease in arm B were allowed to crossover to arm D at the discretion of the treating physician.
Arm/Group | B: Pomalidomide and Dexamethasone | C: Pomalidomide, Dexamethasone, Cyclophosphamide | D: Crossover Arm
Number analyzed (Participants) | 35 | 33 | 17
percentage of participants
  Anemia | 11.4 | 24.2 | 5.9
  Febrile neutropenia | 11.4 | 12.1 | 0
  Fatigue | 8.6 | 1.21 | 0
  Flu-like symptoms | 0 | 0 | 5.9
  Lung infection | 11.4 | 9.1 | 5.9
  Sepsis | 0 | 9.1 | 0
  Upper respiratory infection | 0 | 6.1 | 0
  Lymphodemia | 11.4 | 9.1 | 11.8
  Neutropenia | 31.4 | 51.5 | 23.5
  Thrombocytopenia | 5.7 | 15.2 | 0
  Leukopenia | 14.3 | 12.1 | 5.9
  Hyperglycemia | 0 | 6.1 | 0
  Hyponatremia | 0 | 6.1 | 0
  Hypophosphatemia | 0 | 0 | 5.9
  Hypoxia | 0 | 0 | 5.9
  Confusion | 0 | 6.1 | 0
  Pneumonitis | 0 | 9.1 | 0
  Thromboembolic event | 0 | 6.1 | 0

ADVERSE EVENTS:
Time Frame: 4 years, 1 month
Description: All participants assigned to Arms A, B, C, plus Arm D group of participants formerly in Arm B (Arm B occurrences listed under B, Arm D occurrences listed under D).
Groups:
- D: Crossover Arm: Phase II: Participants who crossed over from Arm B to Arm D.
Arm/Group | A: Dose Escalation of Cyclophosphamide | B: Pomalidomide and Dexamethasone | C: Pomalidomide, Dexamethasone, Cyclophosphamide | D: Crossover Arm
Serious Adverse Events (participants affected / at risk) | 10/10 | 11/36 | 19/34 | 9/17
Other Adverse Events (participants affected / at risk) | 10/10 | 35/36 | 33/34 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Dose Escalation of Cyclophosphamide (N=10) | B: Pomalidomide and Dexamethasone (N=36) | C: Pomalidomide, Dexamethasone, Cyclophosphamide (N=34) | D: Crossover Arm (N=17)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 4 (4) | 2 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal vascular disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders, Other (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
General disorders - Other (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 4 (4) | 3 (4) | 3 (3)
Sepsis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorders - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Dose Escalation of Cyclophosphamide (N=10) | B: Pomalidomide and Dexamethasone (N=36) | C: Pomalidomide, Dexamethasone, Cyclophosphamide (N=34) | D: Crossover Arm (N=17)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 15 (21) | 17 (54) | 6 (10)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Blood and Lymphatic System Disorders - Other (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (10) | 16 (36) | 20 (76) | 8 (18)
Platelet count decreased (Investigations) | 8 (10) | 10 (15) | 16 (46) | 2 (2)
White blood cell decreased (Investigations) | 2 (3) | 7 (13) | 8 (52) | 4 (15)
Lymphocyte count decreased (Investigations) | 0 (0) | 4 (20) | 4 (24) | 3 (15)
Weight gain (Investigations) | 0 (0) | 3 (4) | 4 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 2 (2) | 1 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 2 (3)
Weight loss (Investigations) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Carbon monoxide diffusing capacity decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin T increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 12 (12) | 7 (9) | 2 (2)
Pain (General disorders) | 1 (1) | 3 (3) | 10 (14) | 1 (1)
Fever (General disorders) | 3 (5) | 6 (6) | 4 (8) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 4 (5) | 6 (7) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 2 (3) | 7 (12) | 2 (2)
Chills (General disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 2 (3) | 2 (2) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Irritability (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Edema trunk (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (2) | 3 (4) | 5 (7) | 3 (3)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 5 (6) | 3 (4) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 5 (8) | 5 (10) | 1 (1)
Sepsis (Infections and infestations) | 4 (5) | 1 (1) | 5 (5) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 2 (2) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Bronchial infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Rhinitis infective (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 6 (7) | 10 (15) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 6 (9) | 10 (11) | 2 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 8 (9) | 6 (7) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (5) | 3 (3) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (6) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 7 (8) | 5 (5) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 5 (7) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 4 (5) | 4 (5) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5) | 6 (7) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 4 (4) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 4 (7) | 1 (1) | 3 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 2 (2) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (4) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 3 (7) | 0 (0) | 1 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (7) | 3 (3) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 2 (3) | 1 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (6) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (6) | 7 (8) | 1 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3) | 4 (4) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (2) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 6 (8) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (5) | 3 (3) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 3 (3) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Body odor (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 4 (4) | 2 (4) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 2 (4) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (5) | 1 (1)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Personality change (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flashing lights (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intraoperative renal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Phase 2 nature of design may have limited power to detect statistically significant differences in some efficacy outcomes and toxicity measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes